CLINICAL TRIAL: NCT07315425
Title: Investigation of the Acute Effects of Blood Flow Restriction Aerobic Exercise on Hemodynamic Responses and Muscle Oxygen in Patients With Interstitial Lung Disease
Brief Title: Acute Hemodynamic Responses to Blood Flow Restriction Aerobic Exercise in Interstitial Lung Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2025 - 1878
Record Dates: First submitted 2025-11-26; First posted 2026-01-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Lung Disease (ILD)
Keywords: Blood Flow Restriction; Interstitial Lung Disease; Muscle Oxygenation; Aerobic Exercise
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is designed as triple-blind. Patients will not know their group assignment. All patients' assessments and training sessions will be conducted at different places and times. Evaluations and interventions will be performed by different physiotherapists. Patient groups will be coded before statistical analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity Aerobic Exercise Training Group (Active Comparator): Participants will perform the treadmill protocol (5-minute warm-up, 20-minute loading, 5-minute cool-down; intensity 30-39% HRR or 30-39% peak VO₂).
  Interventions: Other: Low-intensity aerobic exercise training
- Blood Flow Restriction (BFR) Low-Intensity Aerobic Exercise Group (Experimental): Participants will perform the treadmill protocol (5-minute warm-up, 20-minute loading, 5-minute cool-down; intensity 30-39% HRR or 30-39% peak VO₂) with the addition of blood flow restriction.
  Interventions: Other: Blood flow restriction (BFR) low-intensity aerobic exercise training

INTERVENTIONS:
Other: Blood flow restriction (BFR) low-intensity aerobic exercise training — Participants will perform a treadmill-based aerobic exercise session at 30-39% of heart rate reserve (HRR) or 30-39% of peak VO₂. The session will consist of 5 minutes of warm-up, 20 minutes of training at target intensity, and 5 minutes of cool-down (total duration: 30 minutes). Before the loading phase begins, a pneumatic external compression device will be placed around both thighs. Blood flow restriction will be applied only during the 20-minute loading phase and will not be used during warm-up or cool-down.
  Arms: Blood Flow Restriction (BFR) Low-Intensity Aerobic Exercise Group
Other: Low-intensity aerobic exercise training — Participants will perform a single supervised aerobic exercise session on a treadmill under physiotherapist supervision. Exercise intensity will be set at 30-39% of heart rate reserve (HRR) or 30-39% of peak VO₂. The protocol will consist of 5 minutes of warm-up, 20 minutes of training at target intensity, and 5 minutes of cool-down (total duration: 30 minutes).
  Arms: Low-intensity Aerobic Exercise Training Group

SUMMARY:
Interstitial lung diseases (ILD)impaired gas exchange and reduced lung elasticity lead to marked reductions in exercise capacity and decreased oxygen consumption due to circulatory limitations. Blood flow restriction (BFR) exercise involves applying external pressure to partially restrict venous return without entirely blocking arterial inflow. This controlled compression induces temporary hypoxic and metabolic stress, triggering high-intensity-like responses that stimulate growth hormone release, increase protein synthesis, and promote muscle hypertrophy. However, the most crucial advantage of blood flow restriction during exercise is its ability to increase muscle mass during aerobic training. IIn individuals with ILD, BFR may offer a safe and practical way to improve muscle mass and exercise capacity with minimal additional strain on the cardiovascular and musculoskeletal systems.Our study aimed to compare the acute effects of low-intensity blood flow restriction aerobic exercise training and low-intensity aerobic exercise training on hemodynamic responses and muscle oxygenation in patients with ILD. Method: 30 patients with a diagnosis of ILD being followed up will be included in the study. Our study was a randomized, crossover, triple-blind, prospective study. Assessments will be performed at the beginning of the study. On the first day, demographic data and clinical findings of the individuals will be collected. Patients will be asked questions, and their responses will be recorded in their medical records. Respiratory function, respiratory muscle strength and endurance, and peripheral muscle strength will be evaluated. 48 hours from the first day, patients' maximal exercise capacity will be assessed with a cardiopulmonary exercise test (CPET), and muscle oxygenation during CPET will be assessed with a Moxy® monitor. Respiratory muscle fatigue will be assessed with an oral pressure monitor before and after the exercise test. The assessments will be completed over two days. One week after the evaluations, patients will be randomly assigned to two groups. One group will receive low-intensity aerobic exercise training, and the other will receive low-intensity aerobic exercise training with blood flow restriction. Muscle oxygenation will be assessed during both exercise sessions, and respiratory muscle fatigue will be measured before and after each session. All participants will receive both exercise sessions.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) constitute a group of disorders that diffusely affect the lungs, causing varying degrees of inflammation, fibrosis, and structural alterations in the lung parenchyma. These diseases may present with either acute or chronic progression and can involve not only the interstitium but also the alveoli, small airways, vascular structures, and pleura. The etiology of ILD is diverse and may be related to identifiable causes such as environmental or occupational exposures, medications, and radiation. Connective tissue diseases-including rheumatoid arthritis, systemic sclerosis, and systemic lupus erythematosus-along with several systemic disorders, may also lead to pulmonary damage and involvement. Systemic diseases can affect the lungs through infections, vasculitis, or inflammatory mechanisms. Globally, approximately two million individuals are affected by ILD, and in Türkiye, the incidence has been reported as 25.8 per 100,000. The most frequently encountered ILD subtypes include sarcoidosis, idiopathic pulmonary fibrosis, and hypersensitivity pneumonitis .

Dyspnea is one of the most common and disabling symptoms in individuals with ILD, substantially reducing quality of life. Respiratory irregularities observed at rest become more pronounced during exercise. Chronic cough is another prevalent symptom in ILD that negatively impacts daily functioning, social interactions, and psychological well-being, and may also indicate disease progression. Impaired gas exchange and reduced lung elasticity lead to a significant decrease in exercise capacity in ILD, resulting in limitations in daily activities. Assessment of exercise capacity is essential for monitoring disease severity and evaluating treatment effectiveness.

In individuals with ILD, progressive circulatory limitations reduce oxygen consumption. Fibrotic changes in the pulmonary vascular bed restrict blood flow, compromising oxygen delivery during exertion and leading to a marked reduction in VO₂ capacity. Pulmonary hypertension and decreased cardiac output further exacerbate this mechanism. During exercise, the oxygen pulse shows limited increase and may plateau or even decrease in some patients. Consequently, heart rate rises disproportionately compared with healthy individuals, increasing peripheral hypoxia and exercise-induced desaturation. Monitoring muscle oxygenation is important for determining how exercise interventions can be optimized to reduce dyspnea and improve exercise capacity.

Blood flow restriction (BFR) exercise was first introduced in 1966; however, it gained more attention in the mid-1980s due to its potential to induce strength gains at low exercise intensities, thereby reducing orthopedic injury risk. The technique relies on applying controlled external pressure to restrict venous return without completely occluding arterial inflow. This results in a temporary hypoxic and metabolically stressful environment distal to the cuff. Accumulation of lactic acid within the ischemic and hypoxic muscle environment leads to a decrease in intramuscular pH. These metabolic stress responses, which are typically observed during high-intensity exercise, stimulate growth hormone release. Growth hormone-mediated IGF-1 secretion enhances protein synthesis within muscle cells, ultimately promoting muscle hypertrophy. A key advantage of restricting blood flow during aerobic exercise is the potential to increase muscle mass even during low-intensity training .

In recent years, the applicability of BFR exercise has been demonstrated across various populations, including older adults, individuals with obesity, and those with cardiovascular conditions. However, most studies have been conducted in athletes and healthy individuals, and research in clinical populations remains limited. For individuals with ILD, BFR training may offer a safe and practical method to enhance both muscle mass and exercise capacity while imposing minimal stress on the cardiovascular and musculoskeletal systems.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of interstitial lung disease according to the European Respiratory Society (ERS) and American Thoracic Society (ATS) diagnostic criteria.
* Willingness to participate in the study and provide written informed consent.

Exclusion Criteria:

* Presence of any acute infection at the time of the study.
* Orthopedic or neurological conditions that may affect exercise capacity.
* Contraindications to exercise testing according to the American College of Sports Medicine (ACSM) guidelines.
* History of COVID-19 infection within the last three months.
* Receiving treatments outside standard medical therapy.
* Presence of peripheral arterial disease.
* Presence of peripheral neuropathy.
* Resting blood pressure greater than 160/100 mmHg.
* History of deep vein thrombosis, pulmonary embolism, or stroke.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Responses | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  The primary outcome of the study will be the acute hemodynamic responses to low-intensity aerobic exercise with and without blood flow restriction in individuals with interstitial lung disease. Heart rate, respiratory rate, systolic and diastolic blood pressure, and peripheral oxygen saturation will be recorded. Maximum heart rate, perceived dyspnea, and fatigue levels reached during the exercise workload will also be documented. Hemodynamic responses will be assessed during two exercise sessions (Session 1 and Session 2), which are separated by a 7-day washout period. Measurements will be obtained before exercise (pre-exercise), during exercise, immediately after exercise, and at the first minute of recovery.
Hemodynamic Responses (Heart Rate) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Heart rate will be measured in beats per minute using a heart rate monitor before exercise, immediately after exercise, and at the first minute of recovery.
Hemodynamic Responses (Systolic Blood Pressure) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Systolic blood pressure will be measured in mmHg using a sphygmomanometer before exercise, immediately after exercise, and at the first minute of recovery.
Hemodynamic Responses (Diastolic Blood Pressure) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Diastolic blood pressure will be measured in mmHg using a sphygmomanometer before exercise, immediately post-exercise, and at the first minute of recovery.
Hemodynamic Responses (Peripheral Oxygen Saturation (SpO₂)) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Oxygen saturation will be recorded using a portable pulse oximeter (SpO₂, %) at baseline, immediately after exercise, and during the first minute of recovery.
Hemodynamic Responses (Respiratory Rate) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Respiratory rate (breaths per minute) will be counted manually or with a monitor before exercise, immediately post-exercise, and at the first minute of recovery.
Hemodynamic Responses (Dyspnea) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Subjective perception of breathlessness will be assessed using the Modified Borg Scale (0-10) before exercise, at peak exercise, immediately after exercise, and at the first minute of recovery. Modified Borg Scale: The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath.
Hemodynamic Responses (Fatigue (Whole-body and Leg)) | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Perceived overall fatigue and leg fatigue will be assessed using the Modified Borg Scale (0-10) at the same time points as dyspnea. Modified Borg Scale: The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means.
Hemodynamic Responses (Maximum Heart Rate) | During the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  The highest heart rate reached during the exercise session will be documented.

SECONDARY OUTCOMES:
Muscle Oxygenation | Pre-exercise and during the exercise test on Day 1, and pre-exercise and during the first and second exercise sessions on Days 2 and 3.
  Muscle oxygenation will be evaluated using the Moxy® muscle oxygen monitor during both cardiopulmonary exercise testing and exercise training sessions. Local muscle oxygen saturation (SmO₂) and total hemoglobin (THb) values will be recorded at rest, immediately after exercise, and at the first minute of recovery.
Maximal Exercise Capacity | Baseline (Day 1)
  Maximal exercise capacity will be evaluated with cardiopulmonary exercise testing (CPET). Breath-by-breath parameters including VO₂ (oxygen consumption, ml/min), VO₂/kg (oxygen consumption per kilogram per minute, ml/min/kg), METs (metabolic equivalents), V̇E (minute ventilation, L/min), V̇CO₂ (carbon dioxide production, ml/min), EqO₂ (ventilatory equivalent for oxygen), EqCO₂ (ventilatory equivalent for carbon dioxide), RER (respiratory exchange ratio), HR (heart rate, beats/min), HRR (heart rate reserve), VO₂/HR (oxygen pulse, ml), RR (respiratory rate, breaths/min), and SpO₂ (oxygen saturation, %) treadmill speed and gradient, and oxygen saturation will be continuously monitored.
Respiratory Muscle Strength | Baseline (Day 1), Days 2 and 3
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using a portable mouth pressure device in accordance with American Thoracic Society and European Respiratory Society guidelines.Respiratory muscle fatigue assessments will be performed before and after exercise testing and repeated before and after each exercise intervention. Baseline assessments represent pre-exercise measurements. Day 2 and Day 3 correspond to the first and second exercise sessions, respectively.
Respiratory Muscle Endurance | Baseline (Day 1)
  Respiratory muscle endurance will be assessed using incremental threshold loading with a Powerbreathe® device.
Peripheral Muscle Strength | Baseline (Day 1), Days 2 and 3
  Quadriceps and shoulder abductor strength will be assessed using a handheld dynamometer. Three measurements will be taken, and the highest value will be recorded. Baseline assessments represent pre-exercise measurements. Day 2 and Day 3 correspond to the first and second exercise sessions, respectively.
Pulmonary function (Forced vital capacity (FVC)) | Baseline (Day 1)
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | Baseline (Day 1)
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | Baseline (Day 1)
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Baseline (Day 1)
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | Baseline (Day 1)
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, peak flow rate (PEF) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak Güçlü, Prof. Dr., Study Director — Gazi University; Şeyma Mutlu Kayaarslan, PT, MSc, Study Chair — Başkent University and Gazi University; Betül Yoleri, PT, MSc, Principal Investigator — Gazi University; Nilgün Yılmaz Demirci, Prof. Dr., Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Freitas EDS, Karabulut M, Bemben MG. The Evolution of Blood Flow Restricted Exercise. Front Physiol. 2021 Dec 2;12:747759. doi: 10.3389/fphys.2021.747759. eCollection 2021. PMID 34925056
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Marti S, Pajares V, Morante F, Ramon MA, Lara J, Ferrer J, Guell MR. Are oxygen-conserving devices effective for correcting exercise hypoxemia? Respir Care. 2013 Oct;58(10):1606-13. doi: 10.4187/respcare.02260. Epub 2013 Mar 19. PMID 23513249
- [Background] Dipla K, Boutou AK, Markopoulou A, Pitsiou G, Papadopoulos S, Chatzikosti A, Stanopoulos I, Zafeiridis A. Exertional Desaturation in Idiopathic Pulmonary Fibrosis: The Role of Oxygen Supplementation in Modifying Cerebral-Skeletal Muscle Oxygenation and Systemic Hemodynamics. Respiration. 2021;100(6):463-475. doi: 10.1159/000514320. Epub 2021 Mar 30. PMID 33784706
- [Background] Degani-Costa LH, Levarge B, Digumarthy SR, Eisman AS, Harris RS, Lewis GD. Pulmonary vascular response patterns during exercise in interstitial lung disease. Eur Respir J. 2015 Sep;46(3):738-49. doi: 10.1183/09031936.00191014. Epub 2015 May 14. PMID 25976688
- [Background] Hansen JE, Wasserman K. Pathophysiology of activity limitation in patients with interstitial lung disease. Chest. 1996 Jun;109(6):1566-76. doi: 10.1378/chest.109.6.1566. PMID 8769513
- [Background] Kozu R, Shingai K, Hanada M, Oikawa M, Nagura H, Ito H, Kitagawa C, Tanaka T. Respiratory Impairment, Limited Activity, and Pulmonary Rehabilitation in Patients with Interstitial Lung Disease. Phys Ther Res. 2021 Apr 1;24(1):9-16. doi: 10.1298/ptr.R0012. eCollection 2021. PMID 33981523
- [Background] Bonini M, Fiorenzano G. Exertional dyspnoea in interstitial lung diseases: the clinical utility of cardiopulmonary exercise testing. Eur Respir Rev. 2017 Feb 21;26(143):160099. doi: 10.1183/16000617.0099-2016. Print 2017 Jan. PMID 28223398
- [Background] Garner J, George PM, Renzoni E. Cough in interstitial lung disease. Pulm Pharmacol Ther. 2015 Dec;35:122-8. doi: 10.1016/j.pupt.2015.10.009. Epub 2015 Nov 3. PMID 26545874
- [Background] Datta D, Normandin E, ZuWallack R. Cardiopulmonary exercise testing in the assessment of exertional dyspnea. Ann Thorac Med. 2015 Apr-Jun;10(2):77-86. doi: 10.4103/1817-1737.151438. PMID 25829957
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Demedts M, Wells AU, Anto JM, Costabel U, Hubbard R, Cullinan P, Slabbynck H, Rizzato G, Poletti V, Verbeken EK, Thomeer MJ, Kokkarinen J, Dalphin JC, Taylor AN. Interstitial lung diseases: an epidemiological overview. Eur Respir J Suppl. 2001 Sep;32:2s-16s. PMID 11816822
- [Background] Tomlinson OW, Markham L, Wollerton RL, Knight BA, Duckworth A, Gibbons MA, Scotton CJ, Williams CA. Validity and repeatability of cardiopulmonary exercise testing in interstitial lung disease. BMC Pulm Med. 2022 Dec 22;22(1):485. doi: 10.1186/s12890-022-02289-0. PMID 36550475
- [Background] Molgat-Seon Y, Schaeffer MR, Ryerson CJ, Guenette JA. Exercise Pathophysiology in Interstitial Lung Disease. Clin Chest Med. 2019 Jun;40(2):405-420. doi: 10.1016/j.ccm.2019.02.011. PMID 31078218
- [Background] Gaunaurd IA, Gomez-Marin OW, Ramos CF, Sol CM, Cohen MI, Cahalin LP, Cardenas DD, Jackson RM. Physical activity and quality of life improvements of patients with idiopathic pulmonary fibrosis completing a pulmonary rehabilitation program. Respir Care. 2014 Dec;59(12):1872-9. doi: 10.4187/respcare.03180. Epub 2014 Sep 2. PMID 25185149
- [Background] Mahler DA, Rosiello RA, Harver A, Lentine T, McGovern JF, Daubenspeck JA. Comparison of clinical dyspnea ratings and psychophysical measurements of respiratory sensation in obstructive airway disease. Am Rev Respir Dis. 1987 Jun;135(6):1229-33. doi: 10.1164/arrd.1987.135.6.1229. PMID 3592398
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Lista-Paz A, Langer D, Barral-Fernandez M, Quintela-Del-Rio A, Gimeno-Santos E, Arbillaga-Etxarri A, Torres-Castro R, Vilaro Casamitjana J, Varas de la Fuente AB, Serrano Veguillas C, Bravo Cortes P, Martin Cortijo C, Garcia Delgado E, Herrero-Cortina B, Valera JL, Fregonezi GAF, Gonzalez Montanez C, Martin-Valero R, Francin-Gallego M, Sanesteban Hermida Y, Gimenez Moolhuyzen E, Alvarez Rivas J, Rios-Cortes AT, Souto-Camba S, Gonzalez-Doniz L. Maximal Respiratory Pressure Reference Equations in Healthy Adults and Cut-off Points for Defining Respiratory Muscle Weakness. Arch Bronconeumol. 2023 Dec;59(12):813-820. doi: 10.1016/j.arbres.2023.08.016. Epub 2023 Sep 29. English, Spanish. PMID 37839949
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Crum EM, O'Connor WJ, Van Loo L, Valckx M, Stannard SR. Validity and reliability of the Moxy oxygen monitor during incremental cycling exercise. Eur J Sport Sci. 2017 Sep;17(8):1037-1043. doi: 10.1080/17461391.2017.1330899. Epub 2017 May 30. PMID 28557670
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] ROUGHTON FJ, FORSTER RE. Relative importance of diffusion and chemical reaction rates in determining rate of exchange of gases in the human lung, with special reference to true diffusing capacity of pulmonary membrane and volume of blood in the lung capillaries. J Appl Physiol. 1957 Sep;11(2):290-302. doi: 10.1152/jappl.1957.11.2.290. No abstract available. PMID 13475180
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Lollgen H, Leyk D. Exercise Testing in Sports Medicine. Dtsch Arztebl Int. 2018 Jun 15;115(24):409-416. doi: 10.3238/arztebl.2018.0409. PMID 29968559
- [Background] Raghu G, Remy-Jardin M, Myers JL, Richeldi L, Ryerson CJ, Lederer DJ, Behr J, Cottin V, Danoff SK, Morell F, Flaherty KR, Wells A, Martinez FJ, Azuma A, Bice TJ, Bouros D, Brown KK, Collard HR, Duggal A, Galvin L, Inoue Y, Jenkins RG, Johkoh T, Kazerooni EA, Kitaichi M, Knight SL, Mansour G, Nicholson AG, Pipavath SNJ, Buendia-Roldan I, Selman M, Travis WD, Walsh S, Wilson KC; American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, and Latin American Thoracic Society. Diagnosis of Idiopathic Pulmonary Fibrosis. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 1;198(5):e44-e68. doi: 10.1164/rccm.201807-1255ST. PMID 30168753
- [Background] Travis WD, Costabel U, Hansell DM, King TE Jr, Lynch DA, Nicholson AG, Ryerson CJ, Ryu JH, Selman M, Wells AU, Behr J, Bouros D, Brown KK, Colby TV, Collard HR, Cordeiro CR, Cottin V, Crestani B, Drent M, Dudden RF, Egan J, Flaherty K, Hogaboam C, Inoue Y, Johkoh T, Kim DS, Kitaichi M, Loyd J, Martinez FJ, Myers J, Protzko S, Raghu G, Richeldi L, Sverzellati N, Swigris J, Valeyre D; ATS/ERS Committee on Idiopathic Interstitial Pneumonias. An official American Thoracic Society/European Respiratory Society statement: Update of the international multidisciplinary classification of the idiopathic interstitial pneumonias. Am J Respir Crit Care Med. 2013 Sep 15;188(6):733-48. doi: 10.1164/rccm.201308-1483ST. PMID 24032382
- [Background] Guler SA, Corte TJ. Interstitial Lung Disease in 2020: A History of Progress. Clin Chest Med. 2021 Jun;42(2):229-239. doi: 10.1016/j.ccm.2021.03.001. PMID 34024399